CLINICAL TRIAL: NCT00384020
Title: Phase 4 Clinical Pharmacogenomics of Antidepressant Response
Brief Title: Clinical Pharmacogenomics of Antidepressant Response
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); Taipei Medical University WanFang Hospital (Other); Taipei City Hospital (Other Government); Mackay Memorial Hospital (Other)
Other Study IDs: MD-095-PP-01; NSC 95-2314-B-400-001
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Depression
Keywords: Major Depression Disorder; Antidepressant; Pharmacogenomics; Cytochrome P450; Serotonin Transporter
MeSH Terms: conditions — Depression | interventions — Paroxetine; Escitalopram

STUDY DESIGN:
Observational Model: Case-Only

INTERVENTIONS:
Drug: Paroxetine (Seroxat)
Drug: Escitalopram (Lexapro)

SUMMARY:
The purpose of this study is to understand how genetic polymorphisms influence the efficacy and side effect profiles of Paroxetine and Escitalopram for major depression treatment.

DETAILED DESCRIPTION:
Despite remarkable progress in recent decades in modern psychopharmacotherapy, patients vary substantially in their response to antidepressants, ranging from total remission to complete treatment failure. Adverse effects, often bothersome and occasionally life-threatening, continue to represent significant challenges to patients and clinicians. Mechanisms responsible for such variability remain poorly understood. In addition, although less appreciated, substantial cross-ethnic variations in psychotropic responses often exist. Recent developments in the field of pharmacogenetics indicate that genetic factors may account for a large part of these differences in response. Specific genetic polymorphisms affecting the function of the serotonin (SERT) system has been postulated to predict the effect of antidepressants. Similarly, genetic mutations have been shown to exert a predominant influence on the expression of a number of drug-metabolizing enzymes, including most of the cytochrome P-450 enzymes that are responsible for the biotransformation of most antidepressants. Polymorphisms of genes controlling these enzymes have been found to be strongly associated with the propensity for various kinds of side effects. Capitalizing on these new developments, the proposed study will examine the predictive value of some of these genetic polymorphisms in 400 patients with DSM-IV major depression prospectively treated with Escitalopram (ECIT) or Paroxetine (PAR). It is postulated that mutations affecting the function of SERT will predict responses to ECIT, polymorphism of CYP2C19 will be associated with the side effect profiles and pharmacokinetics of ECIT.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as of Taiwanese/Chinese ethnic background, and report that both of their parents and all four or three of their grandparents are members of the same ethnic group;
* HAMD-21 > 17 plus MDE (i.e., current major depressive episode) based on SCID;
* male or female, who, if of child-bearing potential, agrees to use effective contraception including the regular use of contraceptive pills, intra-uterine devises or abstinence;
* age >= 18;
* capable of giving informed consent;

Exclusion Criteria:

* diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, schizotypal disorder, psychotic depression, bipolar disorders;
* current drug or alcohol abuse or dependence or history of drug or alcohol abuse or dependence within the past 6 months;
* unstable medical or neurological conditions that are likely to interfere with the treatment of depression;
* history of allergy to antidepressants;
* history of seizure disorder;
* pregnancy;
* active suicidal ideation or other safety issues determined by the clinician to not be suitable for inclusion in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: depressive patients in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keh-Ming Lin, MD, MPH, Study Director — National Health Research Institutes, Taiwan; Chia-Hui Chen, MD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (4):
- Taiwan (4):
  - Song-De Branch, Taipei City Hospital, Taipei, Taipei
  - Municipal Wan Fang Hospital, Taipei, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District, Taoyuan

REFERENCES:
- [Derived] Tsai MH, Lin KM, Hsiao MC, Shen WW, Lu ML, Tang HS, Fang CK, Wu CS, Lu SC, Liu SC, Chen CY, Liu YL. Genetic polymorphisms of cytochrome P450 enzymes influence metabolism of the antidepressant escitalopram and treatment response. Pharmacogenomics. 2010 Apr;11(4):537-46. doi: 10.2217/pgs.09.168. PMID 20350136